CLINICAL TRIAL: NCT04672577
Title: Infection Tracking in Travellers (ITIT)
Brief Title: Infection Tracking in Travellers. The Project Aims to Identify Profiles of Travel-associated Illness and to Follow up on Long-term Sequelae of Arboviral Infections and Malaria
Acronym: ITIT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Patricia Schlagenhauf (Other)
Collaborators: ETH Zurich (Other); Swiss Tropical & Public Health Institute (Other); University Hospital, Geneva (Other); Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Patricia Schlagenhauf, Prof. Dr., University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: ITIT
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Travel-Related Illness; Malaria; Dengue; Chikungunya; Zika; SARS-CoV Infection; MERS; Influenza; Diarrhea
MeSH Terms: conditions — Travel-Related Illness; Malaria; Dengue; Chikungunya Fever; Zika Virus Infection; Severe Acute Respiratory Syndrome; Influenza, Human; Diarrhea | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arboviral infection or malaria positive cohort
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — No intervention is planned

SUMMARY:
The investigators hypothesize that sex, age, area of exposure and purpose of travel are associated with different travel-related infections. The investigators also hypothesize that certain infections will have long-term sequelae.

Health-data will be collected from travellers from Switzerland and Europe. The project starts with a pilot study for 50 travellers, followed by the recruiting of 10,000 travellers. The data collection will be via a mobile App (ITIT). The ITIT App will collect active data from travellers. The participants will download the App after signing an electronic consent form and completing a baseline questionnaire. Then the travellers will answer a short daily questionnaire about illness symptoms during travel. The ITIT App will also collect passive data (GPS localisation, environmental and weather data). The project will provide real-time data on travel-related infections and profile travel illness by age, sex and purpose of travel and also identify outbreaks.

DETAILED DESCRIPTION:
International travel is growing exponentially. Globally, there will be a projected 1.8 billion traveller arrivals in 2030. Current surveillance of travellers' health is top-down (i.e., clinicians/laboratories report illness) and only a small proportion of illness events are captured. More data are needed on the types of infections acquired by different groups who have varying purposes of travel such as business/corporate travellers, those visiting friends and relatives (VFR), leisure/tourist travellers and mass gathering event (Hajj, Olympics, World Cup) attendees. More data are needed to profile infections in travellers according to age and sex as men and women have different infection susceptibilities. Infectious diseases, in particular the spread of malaria and "arboviral infections",(i.e. viruses such as dengue) pose major threats with changing epidemiology influenced by climate, environmental factors and human mobility. The extent and impact of these infections on travellers' health and their long-term sequelae have scarcely been evaluated. The collected data will allow the profiling of infections in travellers according to purpose of travel and according to age and sex. Men and women have different infection susceptibilities but there is just one study on this theme in the context of travel medicine Infectious diseases, in particular the spread of malaria and "arboviral infections", i.e. viruses such as dengue, chikungunya and Zika pose major threats with changing areas of transmission influenced by climate and mobility. Although airline statistics are available on traveller numbers, the volume of ill, returning, possibly viremic travellers entering areas, where susceptible vectors exist has never been quantified. The situation of a twin presence of viremic travellers and competent Aedes vectors may lead to the onward transmission of arboviral infections. The ITIT project, evaluating in-travel and post-travel illness profiles, coupled with geo-location and meteorological data, will yield the granular data needed for personalized travel medicine. This is important given the heterogenicity and increasing volume of global travellers. The project has the support of the World Health Organization (WHO). Since the data will be collected anonymously via a questionnaire on the designed mobile App and the study is non-interventional, the risk category for this project is minimal (A).

ELIGIBILITY:
Inclusion Criteria:

1. travellers who cross international borders
2. adults (over 18 years old)
3. those traveling for more than 2 days and less than 8 weeks

Exclusion Criteria:

1. Non travellers (not crossing international borders)
2. Minors (under 18 years old)
3. those traveling for less than 2 days and longer than 8 weeks

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: International travellers who cross international borders and are traveling for varying purposes such as business/corporate travellers, those visiting friends and relatives (VFR), leisure/tourist travellers and mass gathering events (Hajj, Olympics, World Cup) attendees.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-01-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of travel-related infectious diseases | 8 weeks
  The Likert scale, self-rating of severity is the unit used to evaluate infectious disease symptoms based on 4 health domains (gastrointestinal symptoms, respiratory symptoms, skin infections and rashes, fever, pain and myalgia) combined with the number of travellers reporting symptoms to get the incidence (travelers with illnesses per 100 travellers).

SECONDARY OUTCOMES:
long-term sequelae of arboviral infections and malaria | 1 year
  The quality-of-life scores and health survey SF-12 version scores will be combined to determine the difference in quality of life due to the infections studied.
change in epidemiology of travel-related infectious diseases | 1 year
  Change in incidence of travel related infectious diseases over time (incidence change/time)

CONTACTS AND LOCATIONS:
Locations (1):
- Epidemiology, Biostatistics and Prevention Institute at the University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Farnham A, Blanke U, Stone E, Puhan MA, Hatz C. Travel medicine and mHealth technology: a study using smartphones to collect health data during travel. J Travel Med. 2016 Sep 4;23(6):taw056. doi: 10.1093/jtm/taw056. Print 2016 Jun. PMID 27592821
- [Background] Findlater A, Moineddin R, Kain D, Yang J, Wang X, Lai S, Khan K, Bogoch II. The use of air travel data for predicting dengue importation to China: A modelling study. Travel Med Infect Dis. 2019 Sep-Oct;31:101446. doi: 10.1016/j.tmaid.2019.07.002. Epub 2019 Jul 5. PMID 31284067
- [Background] Leta S, Beyene TJ, De Clercq EM, Amenu K, Kraemer MUG, Revie CW. Global risk mapping for major diseases transmitted by Aedes aegypti and Aedes albopictus. Int J Infect Dis. 2018 Feb;67:25-35. doi: 10.1016/j.ijid.2017.11.026. Epub 2017 Nov 28. PMID 29196275
- [Background] Ponce C, Dolea C. The World Health Organisation (WHO) and International Travel and Health: New collaborative, evidence-based and digital directions. Travel Med Infect Dis. 2019 Jan-Feb;27:1. doi: 10.1016/j.tmaid.2019.01.012. Epub 2019 Jan 17. No abstract available. PMID 30660556
- [Background] Schlagenhauf P, Chen LH, Wilson ME, Freedman DO, Tcheng D, Schwartz E, Pandey P, Weber R, Nadal D, Berger C, von Sonnenburg F, Keystone J, Leder K; GeoSentinel Surveillance Network. Sex and gender differences in travel-associated disease. Clin Infect Dis. 2010 Mar 15;50(6):826-32. doi: 10.1086/650575. PMID 20156059
- [Background] Schlagenhauf P, Tschopp A, Johnson R, Nothdurft HD, Beck B, Schwartz E, Herold M, Krebs B, Veit O, Allwinn R, Steffen R. Tolerability of malaria chemoprophylaxis in non-immune travellers to sub-Saharan Africa: multicentre, randomised, double blind, four arm study. BMJ. 2003 Nov 8;327(7423):1078. doi: 10.1136/bmj.327.7423.1078. PMID 14604928
- [Background] Tomasello D, Schlagenhauf P. Chikungunya and dengue autochthonous cases in Europe, 2007-2012. Travel Med Infect Dis. 2013 Sep-Oct;11(5):274-84. doi: 10.1016/j.tmaid.2013.07.006. Epub 2013 Aug 17. PMID 23962447
- [Derived] Hedrich N, Lovey T, Bernhard J, Grobusch MP, Gautret P, Schlagenhauf P; ITIT Global Network. Real-time illness monitoring in travellers: an international, prospective, digital surveillance study. Travel Med Infect Dis. 2025 Nov-Dec;68:102943. doi: 10.1016/j.tmaid.2025.102943. Epub 2025 Nov 17. PMID 41260318
- [Derived] Lovey T, Hedrich N, Grobusch MP, Bernhard J, Schlagenhauf P; ITIT Global Network. Surveillance of global, travel-related illness using a novel app: a multivariable, cross-sectional study. BMJ Open. 2024 Jul 27;14(7):e083065. doi: 10.1136/bmjopen-2023-083065. PMID 39067885